CLINICAL TRIAL: NCT06749782
Title: Semi-automatic Measurement of Renal Volume at Computed Tomography (CT) Angiography to Plan Repair of Aortic Aneurysms in Patients With Horseshoe Kidney: a Retrospective Study
Brief Title: Semi-automatic Measurement of Renal Volume at CT Angiography to Plan Repair of Aortic Aneurysms in Patients With Horseshoe Kidney.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Antonio Esposito, Professor, IRCCS San Raffaele
Other Study IDs: HR-AAA-CT
Record Dates: First submitted 2024-11-21; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: The Horseshoe Kidney

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: TC — Radiation: Computed Tomography (CT)
  Other Names: Radiation: Computed Tomography (CT)

SUMMARY:
The horseshoe kidney (HK) is a congenital anomaly in which the kidneys are fused in front of the anterior aortic wall in its most common form. The association of abdominal aortic aneurysm (AAA) and horseshoe kidney (HK) is a rare and challenging condition, occurring in less than 0.2% of all AAA cases. In these cases, open surgery is still widely practiced in many centers, with either a transperitoneal or retroperitoneal approach. Typically, several polar arteries arise from the distal abdominal aorta or the iliac arteries to perfuse the HK.

A key consideration for the surgery is whether or not to preserve the vascularization of the variant kidney. Preserving them can be challenging, but removing them can lead to a significant reduction in renal volume and subsequent loss of function. In open surgery repair, it is recommended to reanastomose as many arteries as possible to the prosthesis, even though this introduces additional technical challenges, especially in emergency situations. Computed Tomography Angiography (CTA) is the best diagnostic test for performing a preoperative vascular assessment.

The purpose of the present study is to develop a semi-automated model on preoperative CCTA to measure the volume of parenchyma perfused by each artery to determine whether or not these should be preserved. The model will be validated on post-surgical CCTA in patients with HK treated for AAA.

Customized use of this tool could be a valuable method in surgical decision making, determining which arteries can be made safe during surgery and addressing a rare but complex clinical need.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥18 years old) surgically treated for AAA with HK at San Raffaele Hospital between January 2019 and December 2023, with appropriate pre- and postoperative CTA, pre- and post CT.

Exclusion Criteria:

* Pediatric patients (age <18 years)
* Absence of pre- and postoperative CT images
* Performance of surgery other than open surgery.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients surgically treated for AAA with HK at San Raffaele Hospital between January 2019 and December 2023, with appropriate pre- and post-operative CTA
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
A semi-automatic model to measure renal volume downstream of each HK artery on presurgical CTA.tomographic angiography validated on surgery. | through study completion, an average of 1 month
  Measurement of renal volume perfused by each artery at preoperative computed tomographic angiography validated on surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Davidovic L, Markovic M, Ilic N, Koncar I, Kostic D, Simic D, Tomic I. Repair of abdominal aortic aneurysms in the presence of the horseshoe kidney. Int Angiol. 2011 Dec;30(6):534-40. PMID 22233614
- [Background] De Caridi G, Massara M, Greco M, Mastrojeni C, Serra R, Salomone I, La Spada M. Surgical Treatment of a Voluminous Infrarenal Abdominal Aortic Aneurysm with Horseshoe Kidney: Tips and Tricks. Ann Vasc Dis. 2015;8(4):324-7. doi: 10.3400/avd.cr.15-00083. Epub 2015 Oct 20. PMID 26730260
- [Background] Dorffner R, Thurnher S, Prokesch R, Youssefzadeh S, Holzenbein T, Lammer J. Spiral CT during selective accessory renal artery angiography: assessment of vascular territory before aortic stent-grafting. Cardiovasc Intervent Radiol. 1998 Mar-Apr;21(2):179-82. doi: 10.1007/s002709900239. PMID 9502690
- [Background] O'Hara PJ, Hakaim AG, Hertzer NR, Krajewski LP, Cox GS, Beven EG. Surgical management of aortic aneurysm and coexistent horseshoe kidney: review of a 31-year experience. J Vasc Surg. 1993 May;17(5):940-7. PMID 8487363
- [Background] Crawford ES, Coselli JS, Safi HJ, Martin TD, Pool JL. The impact of renal fusion and ectopia on aortic surgery. J Vasc Surg. 1988 Oct;8(4):375-83. doi: 10.1067/mva.1988.avs0080375. PMID 3172375
- [Background] O'Brien J, Buckley O, Doody O, Ward E, Persaud T, Torreggiani W. Imaging of horseshoe kidneys and their complications. J Med Imaging Radiat Oncol. 2008 Jun;52(3):216-26. doi: 10.1111/j.1440-1673.2008.01950.x. PMID 18477115